CLINICAL TRIAL: NCT06920628
Title: PET Imaging of Cyclooxygenase-1 in Participants With Neurological Manifestations of Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002117; 002117-M
Record Dates: First submitted 2025-04-09; First posted 2025-04-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09-17

CONDITIONS: Long COVID; Post Acute Sequelae of COVID-19
Keywords: Inflammation; COVID; SARS; Neuro-PASC
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Inflammation | interventions — 11C-PS13

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- one arm (Other): All subjects will receive the same tests
  Interventions: Drug: 11C-PS13

INTERVENTIONS:
Drug: 11C-PS13 — Injected IV followed by PET scanning.

SUMMARY:
Background:

SARS-CoV-2 is the virus that causes COVID-19. Some people who recover from COVID-19 have long-term symptoms that affect the brain. These include headaches; loss of taste and smell; sleep problems; thinking problems; depression; and anxiety. Researchers want to know if a tracer (a substance that is injected into a person s body before an imaging scan) can help identify inflammation in people with these brain disorders.

Objective:

To see if a radioactive tracer ([11C]PS13) can highlight brain inflammation in those who had COVID-19 but still have symptoms that affect the brain.

Eligibility:

Adults aged 18 to 70 years with post COVID-19 brain disorders who are enrolled in protocol 000089 or 000711. Healthy volunteers are also needed.

Design:

Participants will have up to 5 clinic visits.

Participants will be screened. They will have blood tests and a test of their heart function.

They will have imaging scans:

Magnetic resonance imaging (MRI): They will lie on a table that slides into a metal tube. Pictures will be taken of the brain.

Positron emission tomography (PET): A needle attached to a thin tube will be inserted into a vein in the arm. The tracer will be injected through the tube. Another needle attached to a thin tube will be inserted into the wrist or inside of the elbow of the other arm to draw blood. They will lie still on a bed while a machine captures images of their brain. The scan will last about 2 hours.

Study involvement is 11 to 14 weeks....

DETAILED DESCRIPTION:
Study Description:

This study will examine whether cyclooxygenase-1 (COX-1), a biomarker of neuroinflammation, is elevated in the brains of individuals with neurological manifestations of Post-Acute Sequelae of SARS-CoV-2 infection (Neuro-PASC).

Objectives:

Primary Objective 1: To determine whether COX-1 is elevated in the striatum of individuals with Neuro-PASC compared to an ageand sex-matched group of healthy volunteers.

Primary Objective 2: To assess the effect of IVIg treatment on Neuro-PASC participants.

Secondary Objective 1: To determine if COX-1 is elevated in all brain regions of individuals with Neuro-PASC compared to healthy volunteers.

Secondary Objective 2: To determine the correlation between COX-1 expression in the striatum of Neuro-PASC participants and three variables: a) plasma CRP levels as an overall measure of inflammation, b) speed on the finger-tapping test, and c) clinical improvement.

Endpoints:

Primary endpoints:

* COX-1 binding in the striatal region (i.e., caudate plus putamen) will be quantified using pharmacokinetic modeling to compare striatal COX-1 in the Neuro-PASC participants to healthy volunteers
* Neuro-PASC participants will be separated into responders and non-responders to the IVIg treatment and scanned a second time to assess COX-1 expression.

Secondary endpoints:

* Comparison of the whole brain COX-1 densities at the voxel level between the Neuro-PASC participants and healthy volunteers.
* COX-1 striatal expression relation to Neuro-PASC participants plasma CRP levels, speed on the finger-tapping test, and clinical improvement.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients: To be eligible for this study, Neuro-PASC participants must meet all of the following criteria:

* Aged 18 to 70 years of age.
* Participants must be in good general health as evidenced by medical history and physical examination.
* Each participant must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
* Participants must have undergone a screening assessment under protocol #000089, Natural History of Post-Coronavirus Disease 19 Convalescence at the National Institutes of Health or #000711 Immunotherapy for Neurological Post-Acute Sequelae of SARSCoV-2 (INPASC) and determined to have neuro-PASC.
* Participants must have had their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Participants must agree to adhere to the lifestyle considerations.

Healthy Volunteers: To be eligible to participate in this study, healthy volunteers must meet all of the following criteria:

* Aged 18 to 70 years of age.
* Able to provide informed consent.
* Be in good general health, as evidenced by medical history and physical examination, and have no cognitive impairment.
* Does not have an active SARS-CoV-2 infection. The protocol will conform with NIH CC standards for documenting a participant does not have active SARS-CoV-2 infection. This may include screening interviews and/or testing.
* Participants must be at least six weeks out since the onset of SARS-CoV-2 symptoms with no fever for at least one week.
* Participants must report having at least one prior SARS-CoV-2 infection.
* Be enrolled in 01M0254, The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers or 17M0181, Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies .
* Have had their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
* Agree to adhere to the lifestyle considerations.

EXCLUSION CRITERIA:

Participants with Neuro-PASC who meet any of the following criteria will be excluded from participation in this study:

* Clinically significant abnormalities on EKG or laboratory testing based on individual clinical judgement. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen). Any lab value that is two times the upper limit or lower values, as per the investigator s judgment. Creatinine level >1.3 mg/dL.
* Participants should not have taken Non-Steroidal Anti-Inflammatory Drug (NSAID)s for two weeks prior to each PET scan. Corticosteroids (with the exception of topical steroids), or immunosuppressants (e.g. methotrexate) must not have been taken within one month prior to each PET scan.
* Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs daily life functions.
* Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
* Are unable to travel to the NIH.
* Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits as determined by the study team.
* Have an inability to lie flat and/or lie still on the camera bed for at least two hours,including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
* Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
* Pregnancy or Breastfeeding Women.
* HIV Infection.

Healthy volunteers who meet any of the following criteria will be excluded from participation in this study:

* Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen).
* Participants should not have taken Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) for two weeks prior to the PET scan. Corticosteroids (with the exception of topical steroids), or immunosuppressants (e.g., methotrexate) must not have been taken within one month prior to the PET scan.
* Participants with an active SARS-CoV-2 infection.
* Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs daily life functions.
* Are unable to travel to the NIH.
* Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
* Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
* Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
* Pregnancy or Breastfeeding Women.
* HIV Infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2028-02-22 (Estimated); Study Completion 2029-02-22 (Estimated)

PRIMARY OUTCOMES:
To measure distribution volume for 11C-PS13 | 36 months
  Target quantification of COX-1

SECONDARY OUTCOMES:
Voxel-wise correlation of distribution volume between healthy volunteers and Neuro-PASC participants | 36 months
  Comparing between COX-1 in healthy volunteers and participants on voxel-level
Correlation of Distribution Volume with CRP | 36 months
  To determine if CRP correlates with COX-1
Correlation of Distribution Volume with Finger Tapping Speed | 36 months
  To determine if Finger-tapping correlates with COX-1
Correlation of Distribution Volume with Clinical Improvement | 36 months
  To determine if Clinical Improvement correlates with COX-1

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The results will be submitted to ClinicalTrials.gov
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol.
Access Criteria: BTRIS

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002117-M.html